CLINICAL TRIAL: NCT01806025
Title: Correlation Between Haptoglobin Phenotypes and Infectious and Other Complications in Cystic Fibrosis Patients
Acronym: Hp-in-CF
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Michal Steinberg, Pulmonology Consultant, Carmel Medical Center
Other Study IDs: CMC-12-0093-CTIL
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Haptoglobin
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Peripheral blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystic Fibrosis Patients: Patients with Cystic Fibrosis with two known severe (class I and class II) mutations
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Cystic Fibrosis is a genetic disease with variable severity, and a predisposition for lung infection. Usually severity is determined by the class of CF mutations, but even among patients with the same severity of mutations there is a variation of the severity of CF.

Haptoglobin has several types (phenotypes), one of them was found to be related to infectious complications.

In this study the investigators aim to find a correlation between Haptoglobin phenotypes in patients with CF and frequency of infectious complications.

To this end the investigators will collect serum from CF patients, and determine their Haptoglobin protein phenotype. The investigators will correlate Haptoglobin phenotype to retrospectively gathered data on infectious complications.

DETAILED DESCRIPTION:
Cystic Fibrosis is a genetic disease with variable severity, and a predisposition for lung infection. The severity of the disease is determined by genetic factors (type of mutation), environmental factors (exposure to bacteria) and behavioral (adherence with therapy). Even among patients with the same severity of mutations there is a variation of the severity of CF.

Haptoglobin is a protein responsible for collecting Iron from senescent Red Blood Cells. There are two genes of Haptoglobin, numbered 1 and 2, and combinations between the two genes create three forms of proteins: 1-1, 1-2, and 2-2. The 1-1 Phenotype was found to be associated with a predisposition to infection.

In this study the investigators aim to find a correlation between Haptoglobin phenotypes in patients with CF and frequency of infectious complications.

To this end the investigators will collect serum from CF patients, and determine their Haptoglobin protein phenotype by gel- electrophoresis. The investigators will correlate Haptoglobin phenotype to retrospectively gathered data on infectious complications.

FEV1- Forced Expiratory Volume in 1 second.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with CF according to diagnostic criteria , between the ages of 0 and 50, who are themselves, or their parents or guardians, able to give informed consent.

Two known severe (class I , II and III) mutations

Exclusion Criteria:

none

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with CF
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
FEV1 | best in last 6 months
  Lung function as determined by spirometry FEV1 (% expected), normalized by age

SECONDARY OUTCOMES:
Number of antibiotic courses per year of follow up | one year
  number of courses of antibiotics the patient received in the last year
Number of days with antibiotics per year of follow up | one year
  number of days the patient received antibiotics
Number Hospitalizations per year | one year
  events of hospitalization
Colonization with bacteria | one year
  colonization of the following bacteria: Pseudomonas aeruginosa (mucoid and non mucoid), Staph aureus (MSSA and MRSA), Hemophilus influenza, Burkholderia Cepacia complex
Presence of CF related diabetes | five years
  presence of CF related diabetes and HbA1C for diabetic patients.

OTHER OUTCOMES:
Haptoglobin phenotype | one visit
  Haptoglobin phenotype in serum will be determined by gel electrophoresis

CONTACTS AND LOCATIONS:
Overall Officials: Michal Shteinberg, MD, Principal Investigator — Pulmonology Institute and CF Center, Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shteinberg M, Rivlin J, Gur M, Konopnicki M, Stein N, Tunney MM, Elborn JS, Downey DG, Johnston E, Shalom H, Levy A. Lack of Association Between Haptoglobin Phenotype and Cystic Fibrosis Outcomes. Lung. 2015 Dec;193(6):1017-21. doi: 10.1007/s00408-015-9801-z. Epub 2015 Sep 14. PMID 26370551